CLINICAL TRIAL: NCT07119749
Title: The Effects of Ingesting Vegan-friendly Whey Protein on Muscle Anabolism and Recovery Following Damaging Eccentric Resistance Exercise
Brief Title: Vegan Whey Protein for Muscle Anabolism and Post-exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RG_21-198
Record Dates: First submitted 2025-05-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Absorptiometry, Photon; Blood Specimen Collection; Resistance Training; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vegan whey protein (Experimental): 3 x daily supplementation of 0.3 g per kg body mass of vegan whey protein isolate for 3 days following an acute bout of lower-body unilateral resistance exercise
  Interventions: Other: Stable isotope tracer consumption; Radiation: DXA scan; Behavioral: Controlled diet; Other: Saliva sample; Other: Blood sample; Procedure: Muscle biopsy; Behavioral: Resistance exercise; Other: Isometric strength test; Dietary Supplement: Supplement
- Dairy whey protein (Active Comparator): 3 x daily supplementation of 0.3 g per kg body mass of dairy whey protein isolate for 3 days following an acute bout of lower-body unilateral resistance exercise
  Interventions: Other: Stable isotope tracer consumption; Radiation: DXA scan; Behavioral: Controlled diet; Other: Saliva sample; Other: Blood sample; Procedure: Muscle biopsy; Behavioral: Resistance exercise; Other: Isometric strength test; Dietary Supplement: Supplement
- Carbohydrate placebo (Placebo Comparator): 3 x daily supplementation of isocaloric carbohydrate placebo for 3 days following an acute bout of lower-body unilateral resistance exercise
  Interventions: Other: Stable isotope tracer consumption; Radiation: DXA scan; Behavioral: Controlled diet; Other: Saliva sample; Other: Blood sample; Procedure: Muscle biopsy; Behavioral: Resistance exercise; Other: Isometric strength test; Dietary Supplement: Supplement

INTERVENTIONS:
Other: Stable isotope tracer consumption — Daily consumption of oral deuterium oxide (0.3 ml per kg of lean body mass) to equilibrate in body water and become slowly incorporated into muscle protein, enabling measurement of muscle protein synthesis rates
Radiation: DXA scan — Whole body DXA scan to assess lean body mass for prescription of deuterium oxide tracer
Behavioral: Controlled diet — Participant will be asked to consume a provided 6-day diet package that will be prepared by the research team. This package will include 3 meals per day plus snacks
Other: Saliva sample — Obtained from participants by asking them to spit into a tube each day during the study, for 11 days in total.
Other: Blood sample — Resting venous blood sample from a forearm vein on 6 separate occasions
Procedure: Muscle biopsy — A highly experienced researcher will sample a small section of muscle (~200 mg) from the vastus lateralis muscle under local anaesthetic (5 ml, 1% Lidocaine)
Behavioral: Resistance exercise — participants will complete 8 sets of 10 repetitions of unilateral eccentric knee extensions on an isokinetic dynamometer.
Other: Isometric strength test — Bilateral isometric strength will be measured using a well-established protocol on an isokinetic dynamometer.
Dietary Supplement: Supplement — Consumption of 3 supplements a day for 3 days following resistance exercise. All supplements are commercially available.

SUMMARY:
This study will be a randomised, double-blind trial where participants will be randomly assigned to consume either a i) vegan whey protein; ii) a whey protein; or iii) a non-protein carbohydrate control supplement for 3 days following strenuous eccentric knee extension exercise. For the duration of the study period, participants will orally consume deuterated water stable isotope tracer (D2O). This, together with repeated blood sampling and muscle biopsies will allow for the calculation of free-living myofibrillar protein synthesis rates under conditions of rest and over 24-, 48- and 72-hours post-exercise recovery.

DETAILED DESCRIPTION:
Participants will be asked to attend 7 experimental visits at the School of Sport, Exercise and Rehabilitation Sciences at the University of Birmingham. The first of the 7 visits will be to assess participant eligibility and to gain written informed consent, where the remaining 6 visits will involve experimental procedures. Briefly, participants will be randomly assigned to ingest one of three nutritional supplements (i: vegan whey protein isolate; ii: whey protein isolate; iii: a non-protein carbohydrate control), 3 times a day for a total of 3 days following an acute bout of unilateral lower-limb eccentric exercise. The study will be run in a double-blinded fashion, where the researchers and participants will both be unaware of nutritional treatment allocation. The amount of protein in each supplemental beverage is prescribed based on total body mass (0.3 g of protein per kg of body mass). As well, for 3 days before and 3 days after the exercise bout, participants will be provided with a standardised diet to consume. For the 3 days before the exercise bout, all participants will consume an identical diet, with a protein intake of 1 g per kg body mass and diets will be energy-matched between treatment groups. For the subsequent 3 days, participants assigned to each of the protein supplementation groups (whey protein or vegan whey protein) will have a daily protein intake of 1.9 g per kg body mass, whereas participants assigned to the carbohydrate control group will maintain protein intake at 1 g per kg body mass. Measures of muscle function, soreness and thickness will be taken before and at various time points after the eccentric exercise, details of which can be found below. To assess the muscle protein synthetic response to each nutritional treatment, participants will orally consume a stable isotope tracer ("heavy water") for a period of 9 days, and muscle biopsies and saliva samples will be taken periodically. An outline of each experimental visit is outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Males, and females aged 18-40 years with a body mass index between 18.5 and 29.9 kg/m2
* Healthy individuals free from metabolic and respiratory disease
* Recreationally active or trained (complete at least 150 mins of moderate physical activity, or 75 mins of vigorous physical activity per week, identify with a certain sport, intend to compete in local competition)
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Demonstrates an understanding of the study and willingness to participate, as evidenced by voluntary written informed consent

Exclusion Criteria:

* Aged <18 or >40 years
* Pregnancy and Breastfeeding
* Body mass index <18.5 or >29.9 kg/m2
* Regular participation (i.e., >3 times weekly for the previous 3 months) in structured exercise or sport with a large eccentric component, such as trail running, soccer, basketball etc.
* Elite athletes or sports-people who compete nationally or internationally
* Habitual smokers
* History of respiratory or metabolic disease
* Any allergies or intolerances to the study materials, protein supplements and food ingredients to be used in this study. In particular, those with an allergy to lidocaine and lactose will be excluded
* Use of any medication or supplements known to affect muscle protein metabolism (e.g., beta-blockers, corticosteroids, analgesics, or non-steroidal anti-inflammatories). Additional medications and/or supplementation aids (e.g., vitamins) will be deemed inappropriate based on the PI's discretion
* Any current or history of musculoskeletal injury
* Any history of medical or surgical events that may affect the study outcomes
* Previous participation in a research-based exercise protocol designed to induce severe muscle damage in the last 6 months
* Habitual protein intakes <0.8 g/kg body mass/day or > 2.2 g/kg body mass/day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis rates (iMyoPS) | 3 days pre-exercise and 3 days post-exercise
  1. Changes in myofibrillar protein synthesis rates of the exercised leg, both over time (1, 24, 48 and 72 hours) during post-exercise recovery and between supplemental groups (vegan whey, whey protein, and non-protein carbohydrate control). Determined by assessing the incorporation of deuterium in muscle, relative to saliva and blood deuterium enrichment.
Muscle function | pre- and 1, 4, 24, 48 and 72 hr post-exercise
  4. Changes in leg muscle architecture followed by leg strength and neural activation will be assessed pre- and at 1, 8-, 24-, 48- and 72-hours post-exercise. Muscle architecture will be assessed using ultrasound and specifically, shear-wave elastography. Change in isometric strength will be assessed on a Biodex dynamometer at a set knee angle while simultaneously assessing neural activation. Participants will be asked to perform a maximal voluntary contraction (MVC) for 5 seconds while neural activation is measured using the interpolated twitch method. There will be 3 measurements for MVC and neural activation with 2 minutes rest between each attempt on visit
Intramuscular anabolic signalling | pre- and 1-hr and 24-hr post-exercise
  2. Changes in the total protein content and phosphorylation status of key anabolic signalling proteins, both over time post-exercise and between the supplemental groups. Assessed by Western Blotting of muscle biopsy samples
Muscle morphology | pre- and 1, 24, 48 and 72 hr post-exercise
  3. Changes in muscle structure and morphology at pre- and at 1, 24-, 48- and 72-hours post-exercise will be assessed via immunofluorescence microscopy of muscle biopsy samples.

SECONDARY OUTCOMES:
Muscle soreness | pre- and 1, 4, 24, 48 and 72 hr post-exercise
  Subjective ratings of muscle soreness will be measured via completion of validated visual analogue scales (no muscle soreness 0 - worst imaginable muscle soreness 100 mm)
Blood markers of muscle damage | pre- and 1, 4, 24, 48 and 72 hr post-exercise
  Plasma concentrations of systemic markers of muscle damage (creatine kinase, lactate dehydrogenase etc) will be measured from blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No